CLINICAL TRIAL: NCT00791999
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Pharmacokinetics and Safety of CDP870 as add-on Medication to MTX in Japanese Active RA Patients Who Have an Incomplete Response to MTX.
Brief Title: Efficacy Confirmation Trial of CDP870 as add-on Medication to Methotrexate (MTX) in Japanese Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDP870-275-08-001; JapicCTI-080665 (Other: JAPIC)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CDP870 100mg (Experimental): 200mg CDP870 given at Week0, 2, 4 and thereafter 100mg CDP870 given every 2 weeks
  Interventions: Drug: CDP870 100mg
- CDP870 200mg (Experimental): 400mg CDP870 given at Week0, 2, 4 and thereafter 200mg CDP870 given every 2 weeks
  Interventions: Drug: CDP870 200mg
- CDP870 400mg (Experimental): 400mg CDP870 given every 2 weeks
  Interventions: Drug: CDP870 400mg
- Placebo (Placebo Comparator): Placebo given every 2 weeks
  Interventions: Drug: Placebo of CDP870

INTERVENTIONS:
Drug: CDP870 400mg — 400mg CDP870 given every 2 weeks until Week22 (SC)
  Arms: CDP870 400mg
Drug: CDP870 200mg — 400mg CDP870 given at Week0, 2, 4 and thereafter 200mg CDP870 given every 2 weeks until Week22 (SC)
  Arms: CDP870 200mg
Drug: CDP870 100mg — 200mg CDP870 given at Week0, 2, 4 and thereafter 100mg CDP870 given every 2 weeks until Week22 subcutaneously(SC)
  Arms: CDP870 100mg
Drug: Placebo of CDP870 — given every 2 weeks until Week22 (SC)
  Arms: Placebo

SUMMARY:
The objective of this trial is to investigate the efficacy (American College of Rheumatology 20% : ACR20) superiority of two dose regiments of CDP870 versus placebo in combination with MTX in active RA patients who have an incomplete response to MTX. The pharmacokinetics and immunogenicity profile of CDP870 will also be investigated to assess the extrapolability of foreign data to the Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of adult-onset RA of at least 6 months but not longer than 15 years in duration as defined by the 1987 American College of Rheumatology classification criteria.
* Subjects must have active RA disease as defined by:

  * At least 9 tender joints and 9 swollen joints
  * ESR of 30 mm/hour or CRP of 1.5 mg/dL
* Subjects must have received treatment with MTX for at least 6 months prior to the start of study drug administration. The dose of MTX must have remain fixed for at least 2 months prior to the study and the dose of MTX should be within 6 to 8 mg/week.

Exclusion Criteria:

* Patients who have a diagnosis of any other inflammatory arthritis
* Patients who have a secondary, non-inflammatory type of arthritis (eg, osteoarthritis, fibromyalgia)
* Patients who currently have, or who have a history of, a demyelinating or convulsive disease of the central nervous system (eg, multiple sclerosis, epilepsy)
* Patients who have NYHA (New York Heart Association) Class III or IV congestive heart failure
* Patients who currently have, or who have a history of, tuberculosis
* Patients who have a high risk of infection (with a current infectious disease, a chronic infectious disease, a history of serious infectious disease)
* Patients who currently have, or who have a history of, malignancy
* Female patients who are breastfeeding or pregnant, who are of childbearing potential
* Patients who previously received treatment with 2 or more anti-TNFα drugs or who previously failed to respond to treatment with 1 or more aint-TNFα drugs.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Chair — OPCJ
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushuh Region
  - Shikoku Region
  - Tohoku Region

REFERENCES:
- [Derived] Yamamoto K, Takeuchi T, Yamanaka H, Ishiguro N, Tanaka Y, Eguchi K, Watanabe A, Origasa H, Shoji T, Sakamaki Y, van der Heijde D, Miyasaka N, Koike T. Efficacy and safety of certolizumab pegol plus methotrexate in Japanese rheumatoid arthritis patients with an inadequate response to methotrexate: the J-RAPID randomized, placebo-controlled trial. Mod Rheumatol. 2014 Sep;24(5):715-24. doi: 10.3109/14397595.2013.864224. Epub 2013 Dec 9. PMID 24313916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Japan between 2008 and 2010.
Pre-assignment Details: Participant flow results are based on the safety set.
Period: Overall Study
Arm/Group | CDP870 100mg | CDP870 200mg | CDP870 400mg | Placebo
Started | 72 | 82 | 85 | 77
Completed | 51 | 66 | 65 | 25
Not Completed | 21 | 16 | 20 | 52
Not completed — Protocol planed withdrawal | 14 | 11 | 11 | 45
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 3 | 0 | 1 | 0
Not completed — Adverse Event | 3 | 3 | 7 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 2
Not completed — Reason other than those above | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDP870 100mg | CDP870 200mg | CDP870 400mg | Placebo | Total
Number analyzed (Participants) | 72 | 82 | 85 | 77 | 316
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 61 | 77 | 66 | 68 | 272
  >=65 years | 11 | 5 | 19 | 9 | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.6) | 50.6 (11.4) | 55.4 (10.3) | 51.9 (11.1) | 53.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 69 | 69 | 66 | 262
  Male | 14 | 13 | 16 | 11 | 54
Region of Enrollment [Number; unit: participants]
  Japan | 72 | 82 | 85 | 77 | 316

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1)Health Assessment Questionnaire-Disability Index (HAQ-DI), 2)C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
Time Frame: Baseline, Week 12
Population: All 316 subjects (72 CDP 100 mg, 82 CDP 200 mg, 85 CDP 100 mg, 77 Placebo) included in the Full Analysis Set (FAS) are included in this analysis
Measure: Number; unit: percentage of participants
Arm/Group | CDP870 100mg | CDP870 200mg | CDP870 400mg | Placebo
Number analyzed (Participants) | 72 | 82 | 85 | 77
percentage of participants | 62.5 | 76.8 | 77.6 | 28.6
Statistical Analysis 1: Comparison: CDP870 100mg vs CDP870 200mg vs CDP870 400mg; For ACR20 responder rate at Week 12, treatment comparisons versus placebo for the two CDP870 dose groups, the CDP870 200 mg group the CDP870 400 mg, were performed. The ACR20 responder rate in the CDP870 100 mg group was used for the secondary analysis; Test type: Superiority or Other; p < 0.025, Regression, Logistic — Wald p-values(vs. placebo) for the comparison of the treatment groups have been calculated using logistic regression with factors for treatment

2. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CDP870 100mg | CDP870 200mg | CDP870 400mg | Placebo
Number analyzed (Participants) | 72 | 82 | 85 | 77
percentage of participants | 61.1 | 73.2 | 71.8 | 24.7
Statistical Analysis 1: Comparison: CDP870 100mg vs CDP870 200mg vs CDP870 400mg vs Placebo; Test type: Superiority or Other; p < 0.05, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 24-week double blind phase, from Baseline to Week 24
Description: Of the 316 subjects in the Full Analysis Set (FAS), 316 are included in the adverse event reporting based upon the Safety Set (SS) population. The Safety Set includes all subjects randomized who received at least 1 dosing.
Arm/Group | CDP870 100mg | CDP870 200mg | CDP870 400mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/72 | 4/82 | 5/85 | 1/77
Other Adverse Events (participants affected / at risk) | 39/72 | 44/82 | 41/85 | 30/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 100mg (N=72) | CDP870 200mg (N=82) | CDP870 400mg (N=85) | Placebo (N=77)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal perforation (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis noninfective (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 100mg (N=72) | CDP870 200mg (N=82) | CDP870 400mg (N=85) | Placebo (N=77)
Conjunctivitis allergic (Eye disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 2 (2)
Administration site reaction (General disorders) | 3 (7) | 1 (1) | 2 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 8 (8) | 3 (3) | 5 (5) | 4 (4)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (8) | 11 (15) | 13 (18) | 9 (10)
Pharyngitis (Infections and infestations) | 5 (5) | 5 (5) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 3 (4) | 3 (3)
Cell marker increased (Investigations) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (2) | 9 (9)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 4 (4) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No